CLINICAL TRIAL: NCT04483544
Title: Immunotherapy in Combination With PARP Inhibition in Advanced Cervical Cancer Patients Functionally Competent or Deficient for the Fanconi Anemia Repair Pathway
Brief Title: Pembrolizumab and Olaparib in Cervical Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual related to change in standard of care treatment for this population.
Sponsor: Baptist Health South Florida (Other)
Collaborators: Florida Department of Health (Other Government); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-JEK-DIA-001
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Results first posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer; Cervical Carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — pembrolizumab; olaparib

STUDY DESIGN:
Intervention Model Description: PD-1 inhibitor pembrolizumab, in combination with the PARP inhibitor olaparib
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): PD-1 inhibitor pembrolizumab, in combination with the PARP inhibitor olaparib
  Interventions: Drug: pembrolizumab; Drug: olaparib

INTERVENTIONS:
Drug: pembrolizumab — PD-1 inhibitor pembrolizumab, 200mg intravenously (IV) every 3 weeks
Drug: olaparib — PARP inhibitor olaparib 300 mg orally, twice daily (BID)

SUMMARY:
The study is a non-randomized, open-label phase II clinical trial to test the investigational combination of the drug pembrolizumab with the drug olaparib in patients diagnosed with advanced or recurrent cervical carcinoma after standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of cervical carcinoma will be enrolled in this study.
2. Cervical cancer is a disease of the female genital tract. No male patients will be enrolled.
3. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
4. Participant must have recurrent cervical cancer and have a low potential for cure with radiation therapy or surgery alone and:

   a. May have received up to 2 prior chemotherapy regimens. Platinum sensitizing agents for radiation therapy are considered a chemotherapy regimen.
5. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and this protocol.
6. Have measurable disease based on RECIST 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
7. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue.
8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed prior to the first dose of treatment.
9. Patient's life expectancy ≥ 16 weeks.
10. Have adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study treatment. Before patients can be enrolled, they must have normal laboratory values as outlined in Table 1. Labs must also fall within normal limits prior to infusion.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to the first dose of treatment (see Appendix 3). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.
3. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
4. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to the first dose of treatment.
5. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
6. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
7. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
8. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
9. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
10. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
11. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
12. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for ≥5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma.
13. Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.

    Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days.
14. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients, or patients with a known hypersensitivity to olaparib or any of the excipients of the product.
15. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
16. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
17. Has an active infection requiring systemic therapy.
18. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV), solid organ, and hematopoietic transplant patients.
19. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.
20. Has a known history of active TB (Bacillus Tuberculosis).
21. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

    Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that interferes with the requirements of the trial or prohibits obtaining informed consent.
22. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
23. Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
24. Has had an allogenic tissue/solid organ/bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
25. Resting ECG and EKG indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (eg., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
26. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) V. 5.0 grade 2) caused by previous cancer therapy, excluding alopecia.
27. Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of Myelodysplastic syndromes and acute myeloid leukemia (MDS/AML).
28. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
29. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cervical cancer is a disease of the female genital tract. No male patients will be enrolled.
Enrollment: 8 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Diaz, MD, Principal Investigator — Miami Cancer Institute at Baptist Health Inc.
Locations (2):
- United States (2):
  - Miami Cancer Institute, Miami, Florida
  - Miami Cancer Institute at Plantation, Plantation, Florida

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make it available

REFERENCES:
- See also: Miami Cancer Institute — https://baptisthealth.net/cancer-care/home

RESULTS

PARTICIPANT FLOW:
Period: Screening
Arm/Group | Treatment
Started | 8
Completed | 8
Not Completed | 0
Period: Treatment (Completed 1 or More Cycles)
Arm/Group | Treatment
Started | 8
Completed | 7
Not Completed | 1
Not completed — Death | 1
Period: End of Treatment
Arm/Group | Treatment
Started | 7
Completed | 7
Not Completed | 0
Period: Post-Treatment
Arm/Group | Treatment
Started | 7
Completed | 2
Not Completed | 5
Not completed — Admitted to hospice | 2
Not completed — Study terminated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Immune Overall Response Rate
Description: Overall objective Response Rate by Immune Response Evaluation Criteria in Solid Tumors (iRECIST) criteria (iORR)
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | Treatment
Number analyzed (Participants) | 8
percent of participants | 16.7 [8.8 to 19.1]

2. Secondary Outcome: Progression Free Survival
Description: Defined among all treated patients as the time from first dose of study drug until the first date of either disease progression or death due to any cause
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 8
months | 4.5 [2.0 to NA] — Upper bound was not reached for time to event analysis due to lack of enough events observed in the study population by the end of follow-up. Specifically, due to small sample size to start, compounded by censoring of data, many patients did not have the event. Therefore, the upper bound of the 95% confidence interval could not be calculated.

3. Secondary Outcome: Number of Patient Reporting Treatment-emergent Adverse Events (TEAEs)
Description: The number of patients reporting treatment emergent adverse events (TEAEs) defined as an AE that occurs or worsens in the period extending from the first dose of study drug to 30 days after the last dose of study drug in this study
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 8
Participants | 8

4. Secondary Outcome: Number of Patients With Baseline Tumor Deficiencies
Description: The number of patients with baseline tumor deficiencies in the Fanconi Anemia pathway associated with antitumor responses to the combination as assessed by the Fanconi Anemia Triple Stain Immunofluorescence assay, performed on archived paraffin embedded tumor tissues.
Time Frame: baseline
Population: The planned Fanconi Anemia Triple Stain Immunofluorescence assay could not be completed due to lack of available resources to conduct the assay.
Arm/Group | Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Duration of Response
Description: Duration of response (DoR), defined as time from documentation of tumor response to disease progression
Time Frame: 3 years
Population: There were not enough data available to analyze duration of response statistically. Only two participants had partial response and none had complete response. Of the two, only one participant had progression so duration of response could be calculated. The other participant did not progress. Duration of response is presented for the one participant.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 1
days | 62 (0)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 6/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=8)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Infections and Infestations - Other, Abscess (Infections and infestations) | 1 (1)
Kidney Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Creatinine Increased (Investigations) | 3 (3)
Platelet Count Decreased (Investigations) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Stroke (Vascular disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=8)
Anemia (Blood and lymphatic system disorders) | 6 (28)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Blurred Vision (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Colonic Obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal Disorders - Other, Hematochezia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (9)
Rectal Ulcer (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (6)
Chills (General disorders) | 1 (1)
Fatigue (General disorders) | 5 (6)
Pain (General disorders) | 1 (2)
Kidney Infection (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 4 (10)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 2 (4)
Creatinine Increased (Investigations) | 3 (7)
Neutrophil Count Decreased (Investigations) | 1 (1)
Platelet Count Decreased (Investigations) | 3 (4)
Thyroid Stimulating Hormone Increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 3 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (13)
Hyponatremia (Metabolism and nutrition disorders) | 3 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flank Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (4)
Urinary Tract Obstruction (Renal and urinary disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and Subcutaneous Disorders - Other, Rash Not Otherwise Specified (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The rapidly evolving field of immunotherapy in cervical cancer moved pembrolizumab to the frontline setting, which made it difficult to recruit eligible participants. The study was terminated early, and statistical analysis could not be completed with the small number accrued. The planned FATSI analysis and correlative studies also were not completed due the collaborating laboratory's closure. With the early termination, a new laboratory was not sought.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT04483544/Prot_SAP_000.pdf